CLINICAL TRIAL: NCT04889911
Title: Development of a Stage-specific Adaptation of a Self-stigma Intervention for People Recovering from a First Episode of Psychosis
Brief Title: Pilot RCT of Self-stigma Treatment for First Episode Psychosis
Acronym: NECT-YA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: John Jay College of Criminal Justice, City University of New York (Other)
Collaborators: Indiana University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: JJayCuny
Record Dates: First submitted 2018-02-23; First posted 2021-05-17 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: First Episode Psychosis; Youth

STUDY DESIGN:
Intervention Model Description: Randomize controlled trial with random assignment to intervention being studied (NECT-YA) or treatment as usual (Coordinated Specialty Care).
Who Masked: Outcomes Assessor
Masking Description: Assessors will be kept blind to participant assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Narrative Enhancement and Cognitive Therapy- Young Adult, Combined with Coordinated Specialty Care (Experimental): NECT is a structured, 20-session group-based treatment called that combines psychoeducation, cognitive restructuring, and elements of narrative psychotherapy. NECT-YA will be modified to meet the needs of people who have experienced an FEP and may have fewer sessions or be provided in individual format or via telehealth for this study. NECT-YA will be offered to participants who are also receiving treatment within Coordinated Specialty Care programs for First Episode Psychosis.
  Interventions: Behavioral: Narrative Enhancement and Cognitive Therapy- Young Adult, Combined with Coordinated Specialty Care; Other: Coordinated Specialty Care
- Coordinated Specialty Care (Active Comparator): Coordinated Specialty Care is an evidence-based treatment for FEP that includes multiple treatment components. The FEP programs in at the recruiting site follow the Coordinated Specialty Care model.
  Interventions: Other: Coordinated Specialty Care

INTERVENTIONS:
Behavioral: Narrative Enhancement and Cognitive Therapy- Young Adult, Combined with Coordinated Specialty Care — NECT is a psychosocial intervention focused on addressing the effects of self-stigma on individuals diagnosed with severe mental illnesses. For the present study, the intervention has been modified to address the needs of youth who have recently experienced a first episode of psychosis.
  Other Names: NECT-YA
  Arms: Narrative Enhancement and Cognitive Therapy- Young Adult, Combined with Coordinated Specialty Care
Other: Coordinated Specialty Care — Coordinated Specialty Care is an evidence-based, multimodal intervention for persons who have experienced a first episode of psychosis.
  Other Names: CSC

SUMMARY:
The overall purpose of the proposed exploratory intervention development application, is to conduct research that will inform the adaptation and preliminary testing of NECT modified for youth (aged 15-24) with first episode psychosis (FEP), targeting self-concept and illness conceptions to increase treatment engagement. The specific aims of the project are to: 1) adapt NECT to be responsive to the needs and preferences of youth with FEP, and 2) Assess the feasibility, acceptability and preliminary effectiveness of the modified intervention (NECT-YA) combined with coordinated specialty care (CSC) services, compared to CSC services alone, in a small (n = 40) RCT.

DETAILED DESCRIPTION:
The investigators will conduct a small RCT of the modified intervention (NECT-YA), combined with CSC, in comparison with CSC alone, with 40 persons recruited from three FEP programs, assessing acceptability and feasibility, and collecting data on primary outcome (service engagement and therapeutic alliance), related outcomes (self-esteem, hopelessness, and social functioning) and mechanisms of action (self-stigma, illness conceptions and coping). The investigators will also collect qualitative data on participants' impressions of NECT-YA, which will inform additional revisions of the manual.

ELIGIBILITY:
Inclusion Criteria:

1. Meets criteria for FEP youth based on the following definition: age 15-24, onset of psychotic symptoms within the last 5 years, and an absence of a primary substance use or mood disorder that could be causing the psychotic symptoms (confirmed by program eligibility);
2. Meets criteria for moderate (defined as a mean score of 1-1.5 on the 0-3 scale of the Internalized Stigma of Mental lllness Scale [ISMI]) or elevated (defined as a mean score of 1.5-3 on the 0-3 scale of the ISMI) self-stigma;
3. Speaks English well enough to complete assessments and participate in groups;
4. Is able to provide informed consent to participate.

Exclusion Criteria:

Does not meet any of the above inclusion criteria.

Ages: 15 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Treatment Engagement | 0 minutes
  Quantity of service use will be measured using attendance records for groups collected by facilitators, as well as administrative data on total service use within the FEP programs.
Working Alliance Inventory Short Form-Client Version | 2 minutes
  A 12-item self-report measure of perception of relationship with the treatment team. Higher scores indicate better working alliance.
Coping with Symptoms Checklist | 15 minutes
  Assesses the use of problem-centered, neutral and avoidant coping strategies to deal with a variety of psychiatric symptoms commonly experienced by people with severe mental illnesses. Higher scores in each subscale indicate more use of that type of coping strategy.

SECONDARY OUTCOMES:
Beck Hopelessness Scale | 3 minutes
  The Beck Hopelessness Scale is a well-established 20-item scale that will be used to measure pessimistic expectations of the future. Individual items are summed to provide an overall index of hope or its absence. Higher scores indicate less hope.
Rosenberg Self Esteem Scale | 2 minutes
  The Rosenberg Self Esteem Schedule will be used to measure self-esteem and self-deprecation. Higher scores indicate more self-esteem.
Quality of Life Scale | 20 minutes
  The Quality of Life Scale is a 21-item scale completed by clinically trained research staff following a semi-structured interview that assesses social functioning in multiple domains. Higher scores indicate great social functioning.

OTHER OUTCOMES:
Internalized Stigma of Mental Illness Scale | 5 minutes
  A 29 item measure of internalized stigma. Higher scores indicate great internalized stigma.
Positive and Negative Syndrome Scale | 20 minutes
  The Positive and Negative Syndrome Scale is a 30-item rating scale of psychiatric symptoms associated with psychosis, completed following a chart review and semi-structured interview. Higher scores indicate more symptoms.
Recovery Style Questionnaire Recovery Style Questionnaire | 5 minutes
  The Recovery Style Questionnaire is a 39 item self-report scale designed to assess the extent to which people with psychosis engage in "sealing over" versus "integration" with regard to how their self-conception.

CONTACTS AND LOCATIONS:
Locations (1):
- Eskenazi Health, PARC Program, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No